CLINICAL TRIAL: NCT03353233
Title: Evaluation of Utility of Ultrasound Guided iPACK Block for Knee Extension After Total Knee Arthroplasty.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00070573
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Knee Osteoarthritis; Primary Total Knee Arthroplasty; Physical Therapy; Pain; Knee Extension
Keywords: iPACK; Interspace between the Popliteal Artery and Capsule of the Knee; Posterior Capsule block; Nerve Block
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Ropivacaine; Dental Occlusion; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- iPACK Block Group (Experimental): A nerve block technique using a numbing medication called ropivacaine.
  Interventions: Drug: Ropivacaine; Procedure: Interspace Between the Popliteal Artery and Capsule of the Knee (iPACK) Block
- Sham Group (Placebo Comparator): The same nerve block technique as above, however using an inactive solution of salt water.
  Interventions: Procedure: Interspace Between the Popliteal Artery and Capsule of the Knee (iPACK) Block; Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — Local anesthetic (numbing drug)
  Other Names: Naropin
  Arms: iPACK Block Group
Procedure: Interspace Between the Popliteal Artery and Capsule of the Knee (iPACK) Block — An ultrasound guided nerve block using a numbing medication called ropivacaine that numbs the nerves to the back of the knee.
  Other Names: iPACK; Posterior Capsule
Drug: Saline — An ultrasound guided nerve block using a medication that does NOT numb the nerve called saline, or salt water.
  Other Names: Salt water placebo
  Arms: Sham Group

SUMMARY:
The purpose of this study is to learn if using an Interspace between the Popliteal Artery and Capsule of the Knee (iPACK) injection technique (also called a "nerve block") that numbs the nerves going to the back part of the knee to aid in physical therapy after surgery. The iPACK technique uses a numbing solution (local anesthetics) that is injected behind the knee to reduce pain and to help straighten the knee. This block may affect movement in the leg and make the legs weak, but thing is rare. A few institutions use the iPACK block for patients having total knee replacements, with the hope of providing good pain relief combined with improved mobility after surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Between 18 and 75 years old
* American Society of Anesthesiologists (ASA) 1-3 patients undergoing primary total knee arthroplasty

Exclusion Criteria:

* ASA 4 or 5
* Revision knee arthroplasty
* Diagnosis of chronic pain
* Daily chronic opioid use (over 3 months of continuous opioid use)
* Inability to communicate pain scores or need for analgesia
* Acute knee dislocation/fracture
* Infection at the site of block placement
* Age under 18 years old or greater than 75 years old
* Pregnant women
* Intolerance/allergy to local anesthetics
* Weight <50 kg
* Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance
* Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; patients will be deidentified and no personal information or medical records used.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iPACK Block Group | Sham Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iPACK Block Group | Sham Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.84 (6.39) | 64.59 (7.01) | 65.71 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 20 | 23 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Able to Hyperextend the Knee After Surgery
Description: Ability to hyperextend the knee after surgery
Time Frame: Within 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | iPACK Block Group | Sham Group
Number analyzed (Participants) | 25 | 25
Participants | 4 | 3

2. Secondary Outcome: Ambulation as Measured by Distance Walked After Surgery
Time Frame: Post-operative Day 0
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | iPACK Block Group | Sham Group
Number analyzed (Participants) | 25 | 25
feet | 120.36 (123.1) | 148.8 (108.4)

3. Secondary Outcome: Pain as Measure by Numerical Rating Scale (NRS) 11
Description: The 11-point numeric rating scale ranges from 0 ("no pain") to 10 ("worst pain imaginable").
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iPACK Block Group | Sham Group
Number analyzed (Participants) | 25 | 25
score on a scale | 4.64 (2.74) | 5 (2.2)

4. Secondary Outcome: Cumulative Opioid Consumption
Description: Total amount of opioids used
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: IV morphine equivalents
Arm/Group | iPACK Block Group | Sham Group
Number analyzed (Participants) | 25 | 25
IV morphine equivalents | 47.52 (39.54) | 48.98 (36.3)

ADVERSE EVENTS:
Time Frame: From enrollment in study until 24 hours post-op.
Arm/Group | iPACK Block Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Technical problems with allocations leading to unrelabile and uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03353233/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03353233/ICF_001.pdf